CLINICAL TRIAL: NCT01676012
Title: High Definition Bronchoscopy; an Exploratory Study of Diagnostic Value in Comparison to Standard White Light Bronchoscopy and Autofluorescence Bronchoscopy
Brief Title: Hd-bronchoscopy, Comparison to Standard White Light and Autofluorescence Bronchoscopy
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 38719
Record Dates: First submitted 2012-08-15; First posted 2012-08-30 (Estimated); Results first posted 2015-05-12 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- five types of bronchoscopy: Bronchoscopy will be performed in a standardized order using five different imaging modes.
  1. Standard white light videobronchoscopy (WLB)
  2. High Definition -Bronchoscopy
  3. HD-bronchoscopy + surface enhancement (iScan-surface)
  4. HD-bronchoscopy + tone enhancement (iScan-tone)
  5. Auto Fluorescence Bronchoscopy (AFB - SAFE3000) in dual video mode

SUMMARY:
Through technological improvement a new technique has become available in the form of high-definition (HD-) bronchoscopy. Current normal video white light bronchoscopy is the standard, and video-autofluorescence bronchoscopy (AFB) is offered by specialized centers only. The impact of this development with high-definition videobronchoscopy using a 1.1 megapixel chip on the diagnostic performance of bronchoscopy is however unknown.

The aim of the present study therefore is to explore the diagnostic performance (sensitivity and specificity) of HD-videobronchoscopy, HD + surface enhancement (iScan filtering technique) and HD + tone enhancement filtering in comparison to standard WLB and dual mode SAFE3000 autofluorescence videobronchoscopy in a high risk population.

DETAILED DESCRIPTION:
Rationale Bronchoscopy is one of the most important procedures in diagnosis of lung cancer and other pulmonary diseases. This procedures renders important anatomical information and subtle changes in the epithelium or vascularity of the bronchial tree are clues to guide the endoscopist in this procedure, especially in case of centrally located lung cancer. These subtle changes may influence the choice of treatment, site of biopsy and resectability of cancers when determining resection margins but also in case of multifocal premalignant disease. A recently published meta-analysis has shown diagnostic superiority of autofluorescence bronchoscopy (AFB) over routine white light bronchoscopy (WLB). Furthermore, patients with a head and neck cancer have an increased risk of developing lung cancer given their smoking habits. Through technological improvement a new technique has become available in the form of high-definition (HD-) bronchoscopy. Current normal video white light bronchoscopy is the standard, and video-autofluorescence bronchoscopy (AFB) is offered by specialized centers only. The impact of this development with high-definition videobronchoscopy using a 1.1 megapixel chip on the diagnostic performance of bronchoscopy is however unknown.

Objective (primary and secondary outcome)

(1) Investigate sensitivity of HD bronchoscopy, with or without surface enhancement or tone enhancement in comparison to AFB (the 'gold standard') and standard WLB for detecting abnormalities of the tracheobronchial tree. Furthermore we aim to investigate determination of resection margins of (suspected) malignancies in the glottic and supraglottic area or centrally located lung cancer in comparison to autofluorescence bronchoscopy (SAFE 3000 dual video mode) in a high risk population with biopsies from all suspect lesions identified by either technique. (2) When the sensitivity and specificity of HD videobronchoscopy in either mode in the abovementioned study is in the vicinity of the reported sensitivity and specificity of SAFE3000 dual mode videobronchoscopy we suggest to use the results of this study perform a power analysis. With this information it may then be possible to design a new future study to compare sensitivity for detecting premalignant lesions in a high risk population in a prospective study.

Study design This study is a descriptive exploratory randomized observational study with a blinded post procedure analysis of the diagnostic performance of HD bronchoscopy in comparison to WLB and AFB.

Study population Patients scheduled for diagnostic or therapeutic procedure under general anesthesia by the cardiothoracic or thoracic surgeon or ear-, nose- and throat (ENT) surgeon with suspected or proven lung cancer or head and neck cancer are eligible for this exploratory study. Eligible are patients with ASA physical status 1-3 patients aged 18 years or older. Ineligibility criteria are all known contraindications for diagnostic bronchoscopy (bleeding disorders, indication for use of anticoagulant therapy (acenocoumarol, warfarins, therapeutic dose of low molecular weight heparins or clopidogrel), known allergy for lidocaine, known pulmonary hypertension, recent and/or uncontrolled cardiac disease). Presence of contraindications for the use of laryngeal mask (anatomical abnormalities, increased risk for intubation (mallampati score 4), ASA classification greater than or equal to 4.

Study procedure Prior to surgery by the ENT surgeon or cardiothoracic surgeon bronchoscopy will be performed by an experienced chest physician through a laryngeal mask under general anaesthesia. Bronchoscopy will be performed in a standardized order using five different imaging modes. The order of the different modes will be randomized. High-definition digital videos will be made from all procedures without in screen indications of date, time or reference to study site or patient identification. The five imaging modes used in this study are: Standard white light videobronchoscopy (WLB); High Definition (HD-) bronchoscopy; HD-bronchoscopy + surface enhancement; HD-bronchoscopy + tone enhancement and Auto Fluorescence Bronchoscopy (AFB - SAFE3000) in dual video mode. All visible abnormalities suspected for malignancy or pre-malignancy will be biopsied afterwards. The HD-digital video's will be reviewed by the experienced bronchoscopists in random order and blinded for patient, study site and date and scored using a predefined scoring system to describe surface, vascularity and tumours. Premalignant lesions identified by multiple techniques are considered as non-inferior. From each patient 5 HD- films will be generated. These films will be reviewed in a blinded fashion and random order by two experienced pulmonologists and an independent equally experienced third pulmonologist. When new clinically relevant abnormalities are found the normally indicated diagnostic procedures will be followed and performed immediately after completion of the videoregistration. All findings will be disclosed to the patient and the physician in charge by the investigator and the impact of these findings on the planned diagnostic or therapeutic procedure will be registered.

Main study parameter / endpoints The bronchoscopy videos will be scored by blinded experienced endoscopists on epithelial changes, vascularity changes, presence or suspicion of dysplasia, presence of suspicion of carcinoma in situ, and tumor margins. The study is a descriptive exploratory study of diagnostic performance of HD-bronchoscopy using different imaging techniques in comparison to standard white light bronchoscopy and autofluorescence bronchoscopy in determining epithelial changes, changes in vascularity and tumour margins. As a secondary outcome we aim, when differences are established between the different bronchoscopy modes, to perform a power analysis to determine the feasibility of a prospectively designed study to investigate the diagnostic performance of HD bronchoscopy.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness After start of the general anaesthesia for the planned operation a laryngeal mask airway is inserted by the anesthesiologist. Bronchoscopy is then performed by a very experienced pulmonologist using routine topical anesthesics. In this way the burden for the patient and the risk of complications is very low. These patients have an indication for the planned surgical procedure and have been evaluated by an anesthesiologist prior to the procedure and are considered fit for surgery. The total anesthesia time for the planned procedure will be increased by 10 to 15 minutes.

Bronchoscopy is a very safe diagnostic procedure, the reported complications are in general attributable to te more invasive diagnostic procedures performed during that diagnostic bronchoscopy like biopsy, lavage and needle aspirations. This is not the aim of this study, invasive diagnostic procedures will only be performed in case of a clinically relevant new finding. In general we expect that the vast majority of the patients involved will not have any benefit of participating in this study

ELIGIBILITY:
Inclusion Criteria:

* Patients fit for surgery and scheduled for diagnostic or therapeutic surgical procedure under general anesthesia by the cardiothoracic or thoracic surgeon or ENT surgeon with suspected or proven lung cancer or head and neck cancer.
* ASA physical status 1-3.
* Age 18 years or older.
* informed consent

Exclusion Criteria:

Contraindications are all known contraindications for diagnostic bronchoscopy such as:

* bleeding disorders,
* indication for use of anticoagulant therapy (acenocoumarol, warfarins, therapeutic dose of low molecular weight heparins or clopidogrel),
* known allergy for lidocaine,
* known pulmonary hypertension,
* recent and/or uncontrolled cardiac disease. Presence of contraindications for the use of laryngeal mask (anatomical abnormalities) increased risk for intubation (mallampati score 4), or compromised upper airway due to extension of primary head and neck cancer.

ASA classification greater than or equal to 4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected or proven head and neck or lung cancer fit for surgery and scheduled for diagnostic or therapeutic surgical procedure in the Radboud University Medical Center Nijmegen
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2012-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: HFM vanderHeijden, MD, Principal Investigator — Principal Investigator
Locations (1):
- Radboud University Medical Center Nijmegen, Nijmegen, Geert Grooteplein 10, Netherlands

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Bronchoscopy will be performed in a standardized order using five different imaging modes.
Groups:
- Five Types of Bronchoscopy: 1. Standard white light videobronchoscopy (WLB)
  2. High Definition -Bronchoscopy
  3. HD-bronchoscopy + surface enhancement (iScan-surface)
  4. HD-bronchoscopy + tone enhancement (iScan-tone)
  5. Auto Fluorescence Bronchoscopy (AFB - SAFE3000) in dual video mode
Period: Overall Study
Arm/Group | Five Types of Bronchoscopy
Started | 32
Completed | 29
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — incomplete set of videos | 1

BASELINE CHARACTERISTICS:
Population: A total of 32 patients were enrolled. Two patients had a insecure airway so bronchoscopy was performed in 30 patients and a complete set of videos was available for analysis in 29 patients.
Arm/Group | Five Types of Bronchoscopy
Number analyzed (Participants) | 29
Age, Continuous [Mean (Full Range); unit: years] | 63 [40 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 18
Region of Enrollment [Number; unit: participants]
  Netherlands | 29

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity
Description: Investigate sensitivity of HD bronchoscopy, with or without surface enhancement or tone enhancement in comparison to AFB (the 'gold standard') and standard WLB for detecting abnormalities of the tracheobronchial tree. So we used 5 types of bronchoscopy; SWL (=standard white light), HD (=high defenition bronchoscopy without surface/tone enhancement), HD-i-Scan1 (=high defention bronchoscopy with surface enhancement), HD-i-scan 2 (=high defenition bronchoscopy with tone enhancement), AFB (=autofluorescence bronchoscopy). Furthermore we aim to investigate determination of resection margins of (suspected) malignancies in the glottic and supraglottic area or centrally located lung cancer in comparison to autofluorescence bronchoscopy (SAFE 3000 dual video mode) in a high risk population with biopsies from all suspect lesions identified by either technique.
Time Frame: one year
Population: Vascular abnormalities were scored most frequently in HD + i-scan2 bronchoscopy. Sites suspicious for preinvasive lesions were most frequently reported using AFB. Tumors were detected equally by all modalities. The preferred modality was HD bronchoscopy with i-scan.
Measure: Mean (Standard Error); unit: # vascular sites detected per patient
Arm/Group | Five Types of Bronchoscopy
Number analyzed (Participants) | 29
# vascular sites detected per patient
  standard white light | 0.28 (0.08)
  HD | 0.72 (0.17)
  HD-i-scan1 | 0.78 (0.22)
  Hd-i-scan2 | 1.33 (0.29)
  AFB | 0.12 (0.05)

2. Secondary Outcome: Sensitivity and Specificity of HD Videobronchoscopy
Description: When the sensitivity and specificity of HD videobronchoscopy in either mode in the abovementioned study is in the vicinity of the reported sensitivity and specificity of SAFE3000 dual mode videobronchoscopy we suggest to use the results of this study perform a power analysis. With this information it may then be possible to design a new future study to compare sensitivity for detecting premalignant lesions in a high risk population in a prospective study.
Time Frame: one year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 11 months
Arm/Group | Five Types of Bronchoscopy
Serious Adverse Events (participants affected / at risk) | 2/29
Other Adverse Events (participants affected / at risk) | 0/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Five Types of Bronchoscopy (N=29)
vocal cord pathology (Respiratory, thoracic and mediastinal disorders) | 1 (1) — After sedation patient was unable to ventilate adequate due to vocal cord pathology. Study procedures were not started.
prolonged hospitalisiation (Respiratory, thoracic and mediastinal disorders) | 1 (1) — After study procedures larynx was lasered. Due to that procedure patient developed oedema wich coused a inspiratory stridor.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No